CLINICAL TRIAL: NCT03953755
Title: Surgery of Secondary Tricuspid Regurgitation
Brief Title: Surgery in Secondary Tricuspid Regurgitation
Acronym: STRONG
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Efremov Sergey, Deputy director for scince, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5/2018
Record Dates: First submitted 2019-05-04; First posted 2019-05-17 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Tricuspid Regurgitation
Keywords: tricuspid regurgitation; tricuspid surgery; moderate tricispid
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control 1 (No Intervention): no/mild tricuspid regurgitation - left-side surgery alone
- moderate TR - left-side surgery (No Intervention): moderate tricuspid regurgitation - left-side surgery alone
- moderate TR - left-side surgery+TVS (Experimental): moderate tricuspid regurgitation - left-side surgery+tricuspid valve surgery
  Interventions: Procedure: Tricuspid valve repair
- Control 2 (No Intervention): tricuspid regurgitation - left-side surgery +tricuspid valve surgery

INTERVENTIONS:
Procedure: Tricuspid valve repair — Tricuspid valve repair
  Arms: moderate TR - left-side surgery+TVS

SUMMARY:
Currently, in cardiology/cardiosurgery the indicators for the surgical correction of secondary tricuspid regurgitationare unclear. AIM: To compare right ventricle structural and functional changes after operation in patients with secondary tricuspid regurgitation with severe mitral /aortic valve pathology, requiring surgical intervention; define the factors influencing major adverse cardiac events depending on the operation/non-operation due to moderate tricuspid regurgitation. This study intends to include 200-300 people and will occur over 5 years with an additional 3-year follow-up.

DETAILED DESCRIPTION:
Background It has been demonstrated in recent large patient monitoring registers that the presence of even mild secondary tricuspid regurgitation (TR) has a significant effect on life expectancy. Currently, in cardiology/cardiosurgery the indicators for the surgical correction of secondary TR are unclear. In this area, international guidelines lack randomized studies and are based on a C level of evidence. C level evidence is based solely on the opinion of experts, retrospective, and/or observational studies. The first indicator for tricuspid valve (TV) surgery is considered to be a combination of TR with severe aortic or mitral valve lesions that require surgical treatment. However, the level of indicators for moderate corrections in such situations is typically II A-B. At the C level of evidence there is no consensus for surgical treatment of such a defect in the international community. Severe TR indicators are Class I while the evidence remains C level because it is not well established that surgical treatment improves the prognosis of these patients. There is a lack of information about the structural and functional changes of the right ventricle after surgery depending on the degree of TR.

Aims and objectives of studying AIM: To compare right ventricle structural and functional changes after operation in patients with secondary tricuspid regurgitation with severe mitral /aortic valve pathology, requiring surgical intervention; define the factors influencing major adverse cardiac events depending on the operation/non-operation due to moderate tricuspid regurgitation.

OBJECTIVES:

1. To study tricuspid regurgitation parameters affecting the long-term prognosis for the surgical correction of severe secondary tricuspid regurgitationof patients with severe aortic/mitral valve pathology requiring surgical treatment.
2. To define hemodynamic parameters of patients with moderate tricuspid regurgitation, when surgical treatment of this defect gives an additional improvement in the short-term and long-term prognosis following surgical treatment of severe aortic/mitral valve diseases.
3. To study changes in contractility parameters in the right ventricle and tricuspid valve function after reconstructive surgery over a period of 3 years.

Methods and study plans This study intends to include 200-300 people and will occur over 5 years with an additional 3-year follow-up.

Inclusion criterion: 1) Signed informed consent form, 2) Previously diagnosed aortic or mitral heart diseases requiring surgical treatment, 3) Over 18 years of age 4) The presence of moderate or severe secondary tricuspid insufficiency.

Exclusion criterion: 1) Significant oncology diseases with a known prognosis of a less than 1 year life expectancy.

Cardiologist examination and survey. Echocardiography All patients will undergo standard echocardiography, including a detailed study of the function and sizes of the right ventricle and right atrium, and measurement of global longitudinal left ventricular deformations using the Speckle Tracking method, peak systolic and diastolic blood flow velocity in TV, fractional changes in area, and tricuspid annulus systolic excursion. Tricuspid regurgitation will be measured according to the standards of EAE/ASE, and will also use the recent 3-tiered classification system of severe insufficiency.

Laboratory techniques Standard for surgical treatment of aortic/mitral valve Coronary catheterization Standard for surgical treatment of aortic/mitral valve, Plan I. Initial visit - cardiologist/cardiosurgeon clinical evaluation - survey and examination II. Echocardiography study - screening - defining degree of tricuspid regurgitation III. Common tests for surgical treatment of aortic/mitral valve IV. Patient randomization with only a moderate degree of TR V. Surgical treatment VI. 30-40 days after surgery - cardiologist examination VII. 90 days after surgery ¬ - cardiologist examination + echocardiography VIII. 1 year after surgery - cardiologist examination + echocardiography IX. 3 years after surgery - cardiologist examination + echocardiography Expected benefits for patients All patients will receive advanced tests using the latest safe ultrasound methods. Frequent echocardiography and patient observations can reveal possible complications after cardiac surgery for aortic/mitral diseases; This study will allow for the correction of drug therapy due to extended diagnosis.

Severe lesions of the tricuspid valve and aortic / mitral heart defects will be corrected in all patients.

New and / or untested methods of treatment will not be used in this study. All surgical procedures will already have undergone testing and been proven effective for the treatment of heart diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Indication left-side valve surgery

Exclusion Criteria:

1. Unwillingness to give informed consent and to enter a regular follow-up program.
2. Prior surgical or percutaneous mitral valve intervention
3. Contraindication to cardiopulmonary bypass (CPB)
4. Clinical signs of cardiogenic shock at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in end-diastolic dimension | 3 month, 1 year, 3 year
  Difference in end-diastolic dimension of right ventricle between of pre- and post- operation
Difference in tricuspid annular plane systolic excursion | 3 month, 1 year, 3 year
  Difference in TAPSE between of pre- and post- operation
Difference in right atrium volume index | 3 month, 1 year, 3 year
  Difference in right atrium volume index between of pre- and post- operation
Difference in fraction of area contraction of right ventricle | 3 month, 1 year, 3 year
  Difference in fraction of area contraction between pre- and post- operation
Difference in right ventricle global strain rate | 3 month, 1 year, 3 year
  Difference in right ventricle global strain rate between of pre- and post- operation
tricuspid regurgitant volume | 3 month, 1 year, 3 year
  tricuspid regurgitant volume
vtricuspid effective regurgitant oriface | 3 month, 1 year, 3 year
  tricuspid effective regurgitant oriface
square of tricuspid regurgitation | 3 month, 1 year, 3 year
  square of tricuspid regurgitation

SECONDARY OUTCOMES:
major adverse cardiac events | 3 month, 1 year, 3 year
  death, myocardial infarction, new hospital readmission, heart transplant, ventricular assist device implantation, aborted sudden death, pulmonary oedema
rate of all-cause death | 3 month, 1 year, 3 year
  all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Shmatov, MD, PhD, Principal Investigator — Saint Petersburg State University, Russia
Locations (1):
- St. Petersburg State University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 year

DOCUMENTS (1):
  • Informed Consent Form (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT03953755/ICF_000.pdf